CLINICAL TRIAL: NCT06519890
Title: Stanford-PIPRA Study: The Accuracy of the Pre-Interventional Preventive Risk Assessment (PIPRA) Tool for the Prediction of ICU-Delirium in a Mixed Cardiothoracic Intensive Care Unit Population
Brief Title: Stanford ICU Delirium PIPRA Study
Acronym: SIDPVS
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jose R Maldonado, MD, Professor of Medicine and Psychiatry, Stanford University
Other Study IDs: IRB #74903
Record Dates: First submitted 2024-03-25; First posted 2024-07-25 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Delirium; Cognitive Impairment; Delirium, Postoperative
Keywords: Artificial Intelligence; Delirium; Delirium Risk Factors; Cognitive Impairment; Postoperative Delirium
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Emergence Delirium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the accuracy of the Pre-Interventional Preventive Risk Assessment (PIPRA) tool in predicting clinical cases of Intensive Care Units (ICU)-delirium, in a population at high risk of developing this syndrome (i.e., admitted patients to Cardiothoracic Intensive Care Units). The population to be studied has already been enrolled in a parallel study intended to determine the accuracy of an electroencephalogram (EEG)-based diagnosis for delirium.

DETAILED DESCRIPTION:
Study investigators would like to determine the real-life accuracy of a new tool developed for the prediction of delirium: Pre-Interventional Preventive Risk Assessment (PIPRA) Tool. The importance of assessing the risk for delirium includes: providing clinicians and patients with accurate predictive information regarding the patient's risk for developing delirium as part of the risk/benefit calculation for surgical procedures and/or admission to an intensive care unit (ICU), and thus potential risk of subsequent cognitive impairment; as well as the ability to introduce timely prophylactic techniques that may prevent its onset.

The PIPRA tools consists of nine items commonly found in any presurgical patient's electronic medical record (EMR). The tool has been designed to run in the background of the EMR and automatically calculate the patient's risk for developing delirium upon admission for surgical intervention. For this study, study investigators will be applying the PIPRA tool to the EMR of patients already enrolled in a parallel study as detailed above.

The PIPRA tool predicts the risk of developing delirium based on its algorithm that takes into consideration the following nine clinical variables: age, height/weight or body mass index, the American Society of Anesthesiologist physical status Classification system (ASA), past history of delirium, past history of cognitive impairment (including dementia), number of medications, preoperative C-reactive protein (CRP) levels, surgical risk (as determined by the European Society of Anesthesiology), and type of surgery. The subsequent result predicts the risk (in percentage) of a patient developing delirium.

The PIPRA tool is fully integrated into EMR systems, operating in the background, extracting relevant information, and automatically generating a delirium prediction score. In addition, this software possesses the flexibility to recalibrate the delirium risk based on the availability of the nine clinical variables.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 18 years or older
2. Clinical suspicion of delirium or subject at risk for delirium 3. Admitted to the Intensive Care Unit (ICU)

4. Expected ICU stay is greater than one (1) day 5. Subject must be fluent in English

Exclusion Criteria:

1. Age is younger than 18 years
2. Subjects with a primary neurological or neurosurgical condition such as stroke, epilepsy, brain tumor, or witnessed seizures, Parkinson's disease, traumatic brain injury, craniectomy, known severe dementia, or Central Nervous System (CNS) infection
3. Active CNS substance abuse, intoxication, or withdrawal
4. Unarousable or unresponsive subjects with Richmond Agitation Sedation Scale (RASS) <-3
5. Subject is blind, deaf, or unable to speak or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stanford Hospital patients requiring admission to the Cardiothoracic ICU
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2024-07-27 (Actual)

PRIMARY OUTCOMES:
Number of subjects with postoperative delirium accurately predicted by the PIPRA Tool | Detection of delirium presenting up to 30 days post-ICU admission
  Assessment of the accuracy on the prediction of subjects identified as developing delirium by the PIPRA tool, as compared with post-operative standardized delirium assessment tools. We will compare the assessment of the PIPRA prediction tool (performed pre-op) with the actual development of delirium as assessed by a clinical assessment based on DSM; the CAM-ICU & SPTD assessment tools.
Development of post-operative Delirium | Up to 30 days post-ICU admission
  Number of subjects diagnosed with post-operative delirium
Development of ICU Delirium | Up to 30 days post-ICU admission
  Number of subjects diagnosed with ICU delirium
Determination of Delirium Phenotype | Up to 30 days post-ICU admission
  For those who develop delirium, the phenotype of delirium will be determined as per the Liptzin-Levkoff Criteria (based on DSM diagnostic Criteria). As such, all delirium episodes will be categorized as: hyperactive, hypoactive, mixed, or subsyndromal delirium.
Sensitivity and specificity of the PIPRA tool for detecting postoperative delirium. | Baseline measurement of variables and detection of delirium presenting up to 30 days post-ICU admission
  Sensitivity and specificity of various cut off points of the PIPRA tool for detecting delirium.
Receiver operating characteristic (ROC) curve analysis of PIPRA tool | Baseline measurement of variables and detection of delirium presenting up to 30 days post-ICU admission
  Receiver operating characteristic (ROC) curve analysis of PIPRA tool

SECONDARY OUTCOMES:
Immediate Postoperative Mortality | From date of ICU admission up to time of discharge from the Intensive Care Unit, an average of two weeks.
  Mortality rate immediately after index surgery
Immediate post-ICU admission Mortality | From date of ICU admission up to time of discharge from the Intensive Care Unit, an average of two weeks.
  Mortality rate following ICU admission
Length of ICU & Hospital Stay | From date of ICU admission up to time of discharge from the ICU, and then from the hospital (assessed up to 1 year after admission)
  Total number of days admitted to the hospital
Discharge Site | Type of facility the patient was discharge to from the hospital (assessed up to 6 months from admission)
  Site of discharge (e.g., home, rehabilitation, skilled nurse facility, etc)
Requirement of Intensive Care Unit Admission | Time to discharge from the hospital (assessed up to 6 months from admission)
  Need for admission to an intensive care unit due to clinical necessity or deterioration
Need of pharmacological protocol | From date of ICU admission up to time of discharge from the ICU (assessed up to 6 months from admission)
  Need of pharmacological agents required for the management of delirium

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Maldonado, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buchan TA, Sadeghirad B, Schmutz N, Goettel N, Foroutan F, Couban R, Mbuagbaw L, Dodsworth BT. Preoperative prognostic factors associated with postoperative delirium in older people undergoing surgery: protocol for a systematic review and individual patient data meta-analysis. Syst Rev. 2020 Nov 14;9(1):261. doi: 10.1186/s13643-020-01518-z. PMID 33189147
- [Result] Dodsworth BT, Reeve K, Falco L, Hueting T, Sadeghirad B, Mbuagbaw L, Goettel N, Schmutz Gelsomino N. Development and validation of an international preoperative risk assessment model for postoperative delirium. Age Ageing. 2023 Jun 1;52(6):afad086. doi: 10.1093/ageing/afad086. PMID 37290122
- [Result] Sadeghirad B, Dodsworth BT, Schmutz Gelsomino N, Goettel N, Spence J, Buchan TA, Crandon HN, Baneshi MR, Pol RA, Brattinga B, Park UJ, Terashima M, Banning LBD, Van Leeuwen BL, Neerland BE, Chuan A, Martinez FT, Van Vugt JLA, Rampersaud YR, Hatakeyama S, Di Stasio E, Milisen K, Van Grootven B, van der Laan L, Thomson Mangnall L, Goodlin SJ, Lungeanu D, Denhaerynck K, Dhakharia V, Sampson EL, Zywiel MG, Falco L, Nguyen AV, Moss SJ, Krewulak KD, Jaworska N, Plotnikoff K, Kotteduwa-Jayawarden S, Sandarage R, Busse JW, Mbuagbaw L. Perioperative Factors Associated With Postoperative Delirium in Patients Undergoing Noncardiac Surgery: An Individual Patient Data Meta-Analysis. JAMA Netw Open. 2023 Oct 2;6(10):e2337239. doi: 10.1001/jamanetworkopen.2023.37239. PMID 37819663
- [Result] Maldonado JR. Acute Brain Failure: Pathophysiology, Diagnosis, Management, and Sequelae of Delirium. Crit Care Clin. 2017 Jul;33(3):461-519. doi: 10.1016/j.ccc.2017.03.013. PMID 28601132
- [Result] Robinson TN, Eiseman B. Postoperative delirium in the elderly: diagnosis and management. Clin Interv Aging. 2008;3(2):351-5. doi: 10.2147/cia.s2759. PMID 18686756